CLINICAL TRIAL: NCT02220803
Title: A Short Term Open, Randomized Cross Over Trial Trial Exploring the Effect of Carbonic Anhydrase Inhibition by Acetazolamide on Sleep Apnea Associated Hypertension
Brief Title: A Short Term Open, Randomized Cross-over Trial Exploring the Effect of Carbonic Anhydrase Inhibition by Acetazolamide on Sleep Apnea Associated Hypertension and Vascular Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Principal Investigator, Jan Hedner, Professor. MD, Göteborg University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CA-BP13; 2013-004866-33 (EudraCT Number)
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Obstructive Sleep Apnea; Sleep-Disordered Breathing; Blood Pressure; Hypertension
Keywords: Acetazolamide; Zonegran; Obstructive Sleep apnea; Apnea; Respiration Disorders; Sleep Disorders; Cardiovascular; Hypertension; Carbonic Anhydrase; Carbonic Anhydrase Inhibitors; Enzyme Inhibitors; Sulfonamides; Therapeutic Uses; Pharmacologic Actions; Vascular stifness
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Hypertension; Apnea; Respiration Disorders; Sleep Wake Disorders | interventions — Acetazolamide; Continuous Positive Airway Pressure

ARMS (3):
- Acetazolamide and CPAP (Active Comparator): Acetazolamide: Diamox®. Hard white capsule, 250 mg. The total treatment is 4 weeks (2+2 weeks). Dosing of acetazolamide will be up-titrated during 3 days according to manufacturer instruction and titration scheme of the study. Maximum dosage (750mg) following titration will be administered as morning (250 mg) and evening(500mg) dosages.Evening medication should be taken 2 hours before bedtime.
  CPAP: Continuous positive nasal airway pressure (nCPAP) delivers slightly pressurized air throughout the breathing cycle and will be given through a mask that is placed and secured over the person's nose. nCPAP titration will follow clinical routines. The standard setting is a pressure delivery in the pressure range 5-15 mbar. The adequate performance of the device is controlled by user time readers and built-in memory cards and control readings are routinely performed at the end of each treatment regimen. Total duration of CPAP treatment is 4(2+2) weeks.
  Interventions: Drug: Acetazolamide; Device: nasal Continuous Positive Airway Pressure (nCPAP)
- CPAP (Active Comparator): Continuous positive nasal airway pressure (nCPAP) delivers slightly pressurized air throughout the breathing cycle and will be given through a mask that is placed and secured over the person's nose. nCPAP titration will follow clinical routines whereby the patient is equipped with an autotitrating device (Sullivan S9). The standard setting is a pressure delivery in the pressure range 5-15 mbar and the full treatment is maintained in the patient´s home. The adequate performance of the device is controlled by user time readers and built-in memory cards and control readings are routinely performed at the end of each treatment regimen. Patients will be encouraged via telephone calls for maximum use. Total duration of CPAP treatment is 4(2+2) weeks.
  Interventions: Device: nasal Continuous Positive Airway Pressure (nCPAP)
- Acetazolamide (Experimental): Acetazolamide (Diamox®) 250 mg. Hard white capsule. The total length of acetazolamide treatment will be 4 weeks (2x2) including 3 days of titration phase of the drug. Dosing of acetazolamide will be up-titrated during 3 days according to manufacturer instruction and titration scheme of the study. Maximum dosage (750mg) following titration will be administered as morning (250 mg) and evening(500mg)dosages.Evening medication should be taken 2 hours before bedtime. The tablets will be swallowed with 300 ml of water (room temperature) in an upright body position and preferably in connection to a meal.
  Interventions: Drug: Acetazolamide

INTERVENTIONS:
Drug: Acetazolamide — Acetazolamide, 250mg tablets, will be administrated as multiple doses. Dosing of acetazolamide will be up-titrated during 3 days according to manufacturer instruction and titration scheme of the study. Maximum daily dosage is 750 mg (equivalent of 3 tablets/daily). Evening medication should be taken 2 hours before bedtime. The total length of Acetazolamide treatment will be 4 weeks (2x2) including 3 days of titration phase of the drug.
  Other Names: Diamox®; ATC-code: S01E C01
  Arms: Acetazolamide; Acetazolamide and CPAP
Device: nasal Continuous Positive Airway Pressure (nCPAP)
  Other Names: nCPAP - Nasal Continuous Positive Airway Pressure.; ResMed - S9 AutoSet™
  Arms: Acetazolamide and CPAP; CPAP

SUMMARY:
This is a short term open, randomized cross over trial to explore and compare the efficacy of pharmacological carbonic anhydrase (CA) inhibition on obstructive sleep apnea (OSA) related hypertension. Patients will be randomized to receive Acetazolamide(Diamox®)(ACZ), Continuous Positive Airway Pressure (CPAP)or CPAP plus ACZ for 2 weeks. Following a 2 week wash-out period all study participants will receive the alternative treatment regimen. The total length of the study will be 10 weeks. The effects of carbonic anhydrase inhibition on blood pressure,hemodynamics and sleep apnea will be investigated.

Study hypothesis:

Carbonic anhydrase inhibition alone or in combination with nCPAP will prominently reduce blood pressure in patients with OSA. Further it is hypothesized that CA inhibition will induce a direct pharmacological effects on vascular stiffness as evidenced in overnight non-invasive assessments of vascular stiffness and that this effect will be particularly strong in patients also responding with a reduction of blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Males 18 to 75 years
* An Apnea-Hypopnea Index (AHI)>15 and an Epworth Sleepiness Scale score (ESS)>6 as verified by a PSG recording.
* Patients with established hypertension (systolic/diastolic blood pressure >= 160/95, either systolic or diastolic accounted for).
* Clinically normal physical findings and laboratory values, as judged by the investigator
* Body mass index >= 35 kg/m2

Exclusion Criteria:

* Hypersensitivity to sulfonamides or acetazolamide-
* Patients with ongoing medication with other sulphonamides or patients any specific antihypertensive treatment.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity.
* Subjects with a seizure disorder
* Patients with clinically verified central sleep apnea
* Clinically significant renal (serum creatinine >2.0 mg/dL or >130 micromol/L), neurological, metabolic (e.g. Type 1 or 2 diabetes), haematological or hepatic disease (ASAT or ALAT >2 times the upper limit of normal).
* Subjects with an occupational risk potentially exaggerated by daytime sleepiness such as handling complex machinery or professional driving
* Unstable angina pectoris, unstable hypertension (or poorly controlled diabetes (HbA1C < 52 mmoles/mol, or fasting plasma glucose >7 mmoles/l).
* Clinically significant congestive heart failure.
* Myocardial infarction or coronary vessel intervention within the previous 6 months period.
* Subjects with uncontrolled hypertension (defined as a diastolic blood pressure ≥110 mmHg and/or a systolic blood pressure ≥180 mmHg with or without medication).
* Previously diagnosed or treated clinically significant cardiac arrhythmia
* Clinically significant chronic pulmonary or gastrointestinal disease.
* Clinical history of depression as judged by the investigator or other previous or present clinically significant psychiatric disease
* Suspected or confirmed poor compliance
* Alcohol or drug abuse during the last year.
* Subjects with any other significant condition that, in the opinion of the investigator, could interfere with participation in the study.
* Severe nocturnal hypoxia defined as more than 10 episodes with an oxygen desaturation exceeding 50% or signs of lacking resaturation between desaturations on previous recordings according to investigators judgment
* Participation in another clinical study during the last 6 months.
* Inability to understand and complete the questionnaires.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is the reduction in systolic/diastolic office blood pressure (mmHg) between the treatment regimens | Baseline to 10 weeks
  The effect will be expressed in terms systolic and diastolic blood pressure (resting office, provoked office and 24 hour).

SECONDARY OUTCOMES:
The secondary objective is to investigate the direct effect of CA inhibition on sleep disordered breathing (Apnea-hypopnea Index, AHI score (events/hour) in the subgroup of patients with OSA after treatment | Baseline to 10 weeks
  Secondary objectives include Apnea-hypopnea Index, AHI score in patients with OSA after treatment.

OTHER OUTCOMES:
Other outcome measures include the assessment of vascular function. | Baseline to 10 weeks
  Vascular function will be assessed by:
  Cold pressor test: assessing vascular response and pulse excitability. Arteriograph: Standard radial pulse assessment to determine pulse wave and augmentation.
  Aritmethic stress test: Evaluate cardiovascular responses such as heart rate, blood pressure and heart rate variability induced by mental work.
  CardioPAT: Finger plethysmograph measuring peripheral arterial tone as well as endothelial function following brachial artery compression (ischemia).
  Full overnight two channel MC Cardio recorder (Sleep apnea indices and recording of continuous oximetry signal for vascular stiffness, microcirculation and chemosensory vascular responsiveness)
  Markers of OSA include:
Markers of OSA such as oxygen desaturation, mean overnight oxygenation, and sleep quality (by polygraphic (PG) assessment, daytime sleepiness, patient-reported outcomes as well as effects on metabolic markers. | Baseline to 10 weeks
  Markers of OSA include: Oxygen desaturation (ODI, events/hour), Mean overnight oxygenation (Spo2, %), Daytime sleepiness: Epworth Sleepiness Scale (ESS), Functional Outcomes of Sleep Questionnaire (FOSQ).
  Patient reported outcomes include: Clinical Global rating Impression and Severity (CGI/S), Columbia suicidal severity rating scale (CSSR-S) Metabolic markers include:Total Cholesterol, HDL, LDL, Triglycerides, Insulin, HbA1C, Fasting plasma glucose and cathecholamines.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hedner, MD. Prof., Principal Investigator — Dept of internal medicine. Center for Sleep and Vigilance disorders.
Locations (1):
- Center for Sleep and Vigilance disorders, Gothenburg, Västra Götaland County, Sweden

REFERENCES:
- [Derived] Eskandari D, Zou D, Grote L, Hoff E, Hedner J. Acetazolamide Reduces Blood Pressure and Sleep-Disordered Breathing in Patients With Hypertension and Obstructive Sleep Apnea: A Randomized Controlled Trial. J Clin Sleep Med. 2018 Mar 15;14(3):309-317. doi: 10.5664/jcsm.6968. PMID 29510792